CLINICAL TRIAL: NCT05406414
Title: Better Sleep Without Medicine - a Cross-sectoral, Quantitative and Qualitative Study for Adult Patients With Mental Disorders and Sleep Problems
Brief Title: The Efficacy of a Transdiagnostic Sleep and Circadian Intervention for Patients With Mental Disorders and Sleep Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADA_1
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-12

CONDITIONS: Depression; Bipolar Affective Disorder; Attention Deficit Disorder
MeSH Terms: conditions — Depression; Bipolar Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic sleep and circadian treatment (Experimental): The intervention group receives sleep treatment consisting of 6 sessions of 60 minutes each over 6 weeks.
  Interventions: Behavioral: Transdiagnostic sleep and circadian treatment
- Active waitlist control group (Active Comparator): The control group receives sleep hygiene education
  Interventions: Behavioral: Active waitlist control group

INTERVENTIONS:
Behavioral: Transdiagnostic sleep and circadian treatment — The intervention group receives sleep treatment consisting of 6 sessions of 60 minutes each over 6 weeks. The sessions are delivered individually and have the following content:
  1. Assessment and introduction to the sleep diary
  2. Review of sleep diary - agreements on behavior changes and goals.
  3. Information on normal sleep, sleep problems and circadian rhythm
  4. Cognitive techniques
  5. Introduction to relaxation training
  6. Follow-up on goals and plan for prevention relapse of sleep problems
  Arms: Transdiagnostic sleep and circadian treatment
Behavioral: Active waitlist control group — The control group receives sleep hygiene education consisting of a single session in which 10 points of sleep advice are presented. They receive a booklet on how to promote good sleep practice and must work on their own for the next 6 weeks to implement this while waiting for the intervention.
  Arms: Active waitlist control group

SUMMARY:
The aim of this study is to examine the effect of a non-pharmacological transdiagnostic sleep intervention as add on to standard treatment for bipolar disorder, depression and attention deficit disorder. Our hypothesis is that the intervention will reduce the severity of the sleep problem and increase sleep quality compared to a control group receiving sleep hygiene education.

DETAILED DESCRIPTION:
Sleep problems include insomnia, circadian rhythm disorders, hypersomnia, and inadequate sleep hygiene. Patients suffering from mental illness are more likely to suffer from sleep problems than the general population. Sleep problems can aggravate the underlying disorder, cause relapse and suicidal ideation. Sleep problems often persist after the mental disorder is successfully treated. Sleep medication is often used but not recommended for long term use. Non-pharmacological treatment of sleep problems is in demand by patients, but treatment options are few. The present intervention is based on a transdiagnostic manual combining Cognitive Behavioral Therapy for Insomnia with chronotherapy, but more research on the efficacy is warranted.

The aim of this study is to investigate whether the intervention reduces the severity of the sleep problem, increases sleep quality, leads to increased sleep efficiency, reduces sleep latency and awakenings, provides better quality of life, increases personal recovery, provides greater readiness to take on a job or reduces consumption of sleep medication.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* F31 Bipolar disorder, F32 unipolar depression or F90 attention deficit disorder
* Insomnia Severity Index (ISI) ≥ 14 (exceeding the threshold for a sleep problem)
* Sleep problems for 3 months: 3 times a week at least one of the following:

  * Sleep onset latency ≥ 30 minutes
  * Wake after sleep onset ≥ 30 minutes
  * Total sleep time ≥ 11 hours per day
  * Displaced circadian rhythm; sleeps earlier than 8 P.M. or later than 02 A.M.
  * Irregular circadian rhythm; bedtime varies ≥ 3 hours throughout the week

Exclusion Criteria:

* Acutely increased suicide risk (Central Regions guideline for assessment of suicide risk)
* Active substance abuse (F10-19)
* The sleep problem can be significantly explained by insufficient treatment of physical
* disease affecting sleep (documented in patients electronic journal)
* Unstable social situation (does not have a permanent residence)
* Shift work (≥ 2 times a week for the last 2 months)
* Pregnancy and breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in the severity of the sleep problem | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint)
  Is measured by Insomnia Severity Index. A self-report instrument measuring the patient's perception of insomnia. The scale ranges from 0 to 28. The higher the score the more severe the insomnia.
Change in sleep quality. | Is measured at inclusion (baseline/ week 0) and at week 6 (endpoint).
  Measured by Pittsburgh Sleeping Quality Index (PSQI). The score is between 0 and 21, "0" indicating no difficulty and "21" indicating severe difficulties.

SECONDARY OUTCOMES:
Change in well-being | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint
  Measured on The WHO-5 Well-Being Index (WHO-5). A questionnaire which measures well-being on a scale ranging from 0 to 100, the higher the score the more well-being.
Level of personal recovery | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint).
  Measured by the questionnaire INSPIRE-O. A questionnaire which measures personal recovery on a scale ranging from 5 to 25, the higher the score the more recovery.
Change in readiness to take on a job | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint)
  Measured by the questionnaire, The Work Ability Index. A score of 0 shows the lowest possibility that the person would take on a job, the score 10 is the highest possibility
Changes in health-related items. | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint)
  The International EQ-5D-5L questionnaire is applied to estimate quality-adjusted years of life.
Change in consumption of sleep medications | Is registered daily during the 6 week study period
  Daily use of sedatives and hypnotics will be measured by medication registration use in sleep diaries during the study period.
Changes in sleep efficiency | Is measured daily during the 6 week study period.
  Is calculated based on the participant's registrations in sleep diaries and by measurements from actigraphs.
Changes in sleep latency | Is measured daily during the 6 week study period
  Is calculated based on the participant's registrations in sleep diaries and by measurements from actigraphs.
Changes in sleep nocturnal awakenings | Is measured daily during the 6 week study period.
  Is calculated based on the participant's registrations in sleep diaries and by measurements from actigraphs.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Kragh, Principal Investigator — Department of affective disorders
Locations (1):
- Mette Kragh, Aarhus C, Denmark

REFERENCES:
- [Derived] Kragh M, Dyrberg H, Speed M, Pedersen P, Kristiansen ST, Martiny K. The efficacy of a transdiagnostic sleep intervention for outpatients with sleep problems and depression, bipolar disorder, or attention deficit disorder: study protocol for a randomized controlled trial. Trials. 2024 Jan 16;25(1):57. doi: 10.1186/s13063-024-07903-6. PMID 38229181